CLINICAL TRIAL: NCT03631030
Title: A Prospective, Single-center, Pilot Study of in Vivo Lesion Characteristics Post Coolief Cooled Radiofrequency Denervation as a Treatment for Chronic Pain
Brief Title: Cooled RF Lesion MRI Characteristics
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: International Spine, Pain and Performance Center (Other)
Collaborators: Halyard Health (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 105-17-0004
Record Dates: First submitted 2018-03-05; First posted 2018-08-15 (Actual); Last update posted 2019-08-07 (Actual); Status verified 2019-08

CONDITIONS: Arthritis;Lumbosacral; Osteo Arthritis Knee; Sacroiliitis; Hip Osteoarthritis; Arthritis, Degenerative
Keywords: Cooled radiofrequency ablation; MRI
MeSH Terms: conditions — Sacroiliitis; Osteoarthritis, Hip; Osteoarthritis

STUDY DESIGN:
Intervention Model Description: Prospective, singe group cohort study
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (1):
- Cooled radiofrequency ablation (Other): This is a single arm study. Patients who will be undergoing cooled radiofrequency ablation for the treatment of arthritis in the cervical facet joints, thoracic facet joints, lumbar facet joints, sacroiliac (SI) region, hip and knee.
  Interventions: Device: Cooled radiofrequency ablation

INTERVENTIONS:
Device: Cooled radiofrequency ablation — Cooled Radiofrequency ablation (CRFA) is a well-established method for delivering lesions into nervous tissue to accomplish neurotomy procedures

SUMMARY:
This Prospective, Single-center, Pilot Study will assist in gaining an understanding of the actual CRFA lesions in an in vivo situation in areas where CRFA is utilized as a standard of care treatment option for the relief of chronic pain (cervical facet joints, thoracic facet joints, lumbar facet joints, Sacroiliac (SI) region, hip and knee).

DETAILED DESCRIPTION:
This study will be a prospective, single-center, pilot study. Adult subjects over the age 21 diagnosed with chronic joint pain (≥ 3 months), scheduled to receive Radiofrequency denervation and meet the selection criteria are eligible to participate in this study. The specific targeted areas of interest in this study will include Cervical facet joints, Thoracic facet joints, Lumbar facet joints, Sacroiliac (SI) region, hip and knee.

The treating physician will follow Standard of Care treatment for all enrolled subjects. As illustrated in Figure 1, the study consists of a screening visit, a treatment visit and a follow up visit. All subjects receiving CRFA will receive an MRI 2 - 7 days after the CRFA procedure. Subjects receiving CRFA of the Sacroiliac Joint will also receive an MRI within 30 days prior to the CRFA procedure. The treating physician may also request an MRI be performed prior to the procedure for subjects receiving CRFA of other targeted areas. The point of enrollment for each subject is the time that they sign the Informed Consent Form.

MRI data will be reviewed by the radiologist on a per patient basis to confirm lesion characteristics. It is anticipated that 3-5 subjects per level will be needed to fully quantify lesion characteristics, however; enrollment will remain flexible for each targeted area based on real time review of MRI data.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥ 21 years
2. Able to understand the informed consent form and provide written informed consent and able to complete outcome measures.
3. Must be clinically appropriate candidate to receive CRFA for treatment of chronic pain.
4. Willing and able to receive an MRI

Exclusion Criteria:

1. Unable to receive an MRI (i.e. due to pacemaker or iron-based metal implant).
2. Unable to receive an MRI (i.e. iron-based metal implant).
3. Extremely thin patients and those with minimal subcutaneous tissue thickness that would not accommodate a radiofrequency lesion of up to 14mm in diameter to limit the risk of skin burns.
4. Active joint infection or systemic or localized infection at the needle entry site (subject may be considered for inclusion once infection is resolved.)
5. Subject currently implanted with a pacemaker or defibrillator
6. In the event a pre-treatment MRI is obtained; trauma or injury occurring to the targeted area between the baseline MRI and CRFA treatment
7. Subject unwillingness or unable to comply with protocol requirements

Min Age: 21 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 15 (Estimated)
Dates: Start 2018-02-25 (Actual); Primary Completion 2020-01 (Estimated); Study Completion 2020-01 (Estimated)

PRIMARY OUTCOMES:
Cooled radiofrequency ablation lesion size | MRI obtained between 2-7 days post-procedure.
  Size in millimeters of cooled radiofrequency ablation lesion via MRI

SECONDARY OUTCOMES:
Pain relief | 2-4 weeks post-procedure as compared to pre-procedure
  Compare pre-procedure and post-procedure change in pain using the numerical pain rating scale with 0 being no pain and 10 being the worst possible pain.

CONTACTS AND LOCATIONS:
Overall Officials: Mehul Desai, MD, MPH, Principal Investigator — International Spine Pain & Performance Center
Locations (2):
- United States (2):
  - International Spine, and Performance Center, Washington D.C., District of Columbia
  - International Spine, Pain and Performance Center, Arlington, Virginia

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Kapural L, Stojanovic M, Sessler DI, Bensitel T, Zovkic P. Cooled radiofrequency (RF) of L5 dorsal ramus for RF denervation of the sacroiliac joint: technical report. Pain Med. 2010 Jan;11(1):53-7. doi: 10.1111/j.1526-4637.2009.00772.x. Epub 2009 Dec 16. PMID 20030745
- [Background] Patel N, Gross A, Brown L, Gekht G. A randomized, placebo-controlled study to assess the efficacy of lateral branch neurotomy for chronic sacroiliac joint pain. Pain Med. 2012 Mar;13(3):383-98. doi: 10.1111/j.1526-4637.2012.01328.x. Epub 2012 Feb 2. PMID 22299761
- [Background] Stelzer W, Aiglesberger M, Stelzer D, Stelzer V. Use of cooled radiofrequency lateral branch neurotomy for the treatment of sacroiliac joint-mediated low back pain: a large case series. Pain Med. 2013 Jan;14(1):29-35. doi: 10.1111/pme.12014. Epub 2012 Dec 28. PMID 23279364
- [Background] Ho KY, Hadi MA, Pasutharnchat K, Tan KH. Cooled radiofrequency denervation for treatment of sacroiliac joint pain: two-year results from 20 cases. J Pain Res. 2013 Jul 4;6:505-11. doi: 10.2147/JPR.S46827. Print 2013. PMID 23869175
- [Background] Kapural L, Mekhail N. Novel intradiscal biacuplasty (IDB) for the treatment of lumbar discogenic pain. Pain Pract. 2007 Jun;7(2):130-4. doi: 10.1111/j.1533-2500.2007.00120.x. PMID 17559482
- [Background] Karaman H, Tufek A, Kavak GO, Kaya S, Yildirim ZB, Uysal E, Celik F. 6-month results of TransDiscal Biacuplasty on patients with discogenic low back pain: preliminary findings. Int J Med Sci. 2010 Dec 14;8(1):1-8. doi: 10.7150/ijms.8.1. PMID 21197258
- [Background] Kapural L, Vrooman B, Sarwar S, Krizanac-Bengez L, Rauck R, Gilmore C, North J, Girgis G, Mekhail N. A randomized, placebo-controlled trial of transdiscal radiofrequency, biacuplasty for treatment of discogenic lower back pain. Pain Med. 2013 Mar;14(3):362-73. doi: 10.1111/pme.12023. Epub 2012 Dec 28. PMID 23279658

DOCUMENTS (2):
  • Study Protocol (2018-05-24): https://cdn.clinicaltrials.gov/large-docs/30/NCT03631030/Prot_000.pdf
  • Informed Consent Form (2018-07-12): https://cdn.clinicaltrials.gov/large-docs/30/NCT03631030/ICF_001.pdf